CLINICAL TRIAL: NCT00691964
Title: A Phase 3, Multi-Center, Randomized, Double-Blind, Placebo-Controlled Study Comparing the Efficacy and Safety of ABT-874 to Etanercept and Placebo in Subjects With Moderate to Severe Chronic Plaque Psoriasis
Brief Title: Study Comparing the Efficacy and Safety of ABT-874 to Etanercept and Placebo in Subjects With Moderate to Severe Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Collaborators: Paragon Biomedical (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M10-114
Record Dates: First submitted 2008-06-04; First posted 2008-06-06 (Estimated); Last update posted 2013-01-21 (Estimated); Status verified 2013-01

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — briakinumab; Etanercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental)
  Interventions: Biological: ABT-874
- B (Active Comparator)
  Interventions: Biological: etanercept
- C (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Biological: ABT-874 — SQ injection 200 mg Weeks 0 and 4; 100 mg Week 8
  Arms: A
Biological: etanercept — SQ injection 50 mg BIW
  Arms: B
Drug: placebo — SQ placebo injections for ABT-874 and etanercept
  Arms: C

SUMMARY:
Compare the efficacy of ABT-874 versus etanercept in subjects with moderate to severe plaque psoriasis

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Psoriasis for 6 mo.
* BSA 10%, PASI 12 or above, PGA 3 or above

Exclusion Criteria:

* Previous exposure to either etanercept or ABT-874

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 347 (Actual)
Dates: Start 2008-05; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who achieve a PGA of 0 or 1 response relative to baseline at Week 12 | 12 Weeks
Proportion of subjects who achieve a PASI 75 response relative to baseline at Week 12 | 12 Weeks

SECONDARY OUTCOMES:
Proportion of subjects who achieve a PASI 100 response relative to baseline at Week 12 | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Martin Kaul, MD, Study Director — AbbVie
Locations (35):
- United States (35):
  - Site Reference ID/Investigator# 8478, Tucson, Arizona
  - Site Reference ID/Investigator# 8462, Fresno, California
  - Site Reference ID/Investigator# 8454, Los Angeles, California
  - Site Reference ID/Investigator# 8476, Denver, Colorado
  - Site Reference ID/Investigator# 9641, Miami, Florida
  - Site Reference ID/Investigator# 8463, Alpharetta, Georgia
  - Site Reference ID/Investigator# 8479, Arlington Heights, Illinois
  - Site Reference ID/Investigator# 8527, Schaumburg, Illinois
  - Site Reference ID/Investigator# 9001, Skokie, Illinois
  - Site Reference ID/Investigator# 8466, West Dundee, Illinois
  - Site Reference ID/Investigator# 8467, Indianapolis, Indiana
  - Site Reference ID/Investigator# 8464, Boston, Massachusetts
  - Site Reference ID/Investigator# 8459, St Louis, Missouri
  - Site Reference ID/Investigator# 8473, East Windsor, New Jersey
  - Site Reference ID/Investigator# 8457, New Brunswick, New Jersey
  - Site Reference ID/Investigator# 8447, Albuquerque, New Mexico
  - Site Reference ID/Investigator# 8475, New York, New York
  - Site Reference ID/Investigator# 8468, Cincinnati, Ohio
  - Site Reference ID/Investigator# 8460, Cleveland, Ohio
  - Site Reference ID/Investigator# 9762, Oklahoma City, Oklahoma
  - Site Reference ID/Investigator# 8480, Lake Oswego, Oregon
  - Site Reference ID/Investigator# 8469, Portland, Oregon
  - Site Reference ID/Investigator# 9566, Portland, Oregon
  - Site Reference ID/Investigator# 9761, Hershey, Pennsylvania
  - Site Reference ID/Investigator# 8471, Philadelphia, Pennsylvania
  - Site Reference ID/Investigator# 8449, Johnston, Rhode Island
  - Site Reference ID/Investigator# 8448, Providence, Rhode Island
  - Site Reference ID/Investigator# 8456, Greer, South Carolina
  - Site Reference ID/Investigator# 8458, Goodlettsville, Tennessee
  - Site Reference ID/Investigator# 8461, Austin, Texas
  - Site Reference ID/Investigator# 10542, Dallas, Texas
  - Site Reference ID/Investigator# 8452, Houston, Texas
  - Site Reference ID/Investigator# 8474, San Antonio, Texas
  - Site Reference ID/Investigator# 8482, Tyler, Texas
  - Site Reference ID/Investigator# 8472, Norfolk, Virginia

REFERENCES:
- [Derived] Gottlieb AB, Leonardi C, Kerdel F, Mehlis S, Olds M, Williams DA. Efficacy and safety of briakinumab vs. etanercept and placebo in patients with moderate to severe chronic plaque psoriasis. Br J Dermatol. 2011 Sep;165(3):652-60. doi: 10.1111/j.1365-2133.2011.10418.x. Epub 2011 Aug 4. PMID 21574983